CLINICAL TRIAL: NCT01212276
Title: A Phase 1 Study of the Safety, Tolerability, Pharmacokinetics and Radiologic Distribution of Ascending Single-Dose Radiolabeled MORAb-028 in Subjects With Metastatic Melanoma
Brief Title: A Safety and MORAb-028 Dose Determination Study in Subjects With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated protocol
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-028-001
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Metastatic Melanoma; Malignant Metastatic Melanoma; Advanced Melanoma; Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): MORAb-028 0.1 mg/kg intravenous
  Interventions: Drug: MORAb-028
- Cohort 2 (Experimental): MORAb-028 0.2 mg/kg intravenous
  Interventions: Drug: MORAb-028
- Cohort 3 (Experimental): MORAb-028 0.5 mg/kg intravenous
  Interventions: Drug: MORAb-028
- Cohort 4 (Experimental): MORAb-028 1.0 mg/kg intravenous
  Interventions: Drug: MORAb-028

INTERVENTIONS:
Drug: MORAb-028 — Cohort 1: 0.1 mg/kg IV on study day 1 only Cohort 2: 0.2 mg/kg IV on study day 1 only Cohort 3: 0.5 mg/kg IV on study day 1 only Cohort 4: 1.0 mg/kg IV on study day 1 only

SUMMARY:
The purpose of this study is to evaluate whether therapy with MORAb-028 is safe, effective, and to determine the appropriate dose of MORAb-028 in the treatment of metastatic melanoma.

DETAILED DESCRIPTION:
Melanoma is a serious form of skin cancer. If untreated, the melanoma can spread beyond the original affected tissue and invade distant tissue and organs. Treatment for metastatic melanoma includes medical treatments (chemotherapy or immunotherapy), surgery, or radiation therapy. MORAb-028 is a recombinant human immunoglobulin M (IgM) monoclonal antibody that recognizes a cell surface diacyl ganglioside named disialoganglioside (GD2). GD2 is overexpressed in tumors of neuro-ectodermal origin such as melanomas, neuroblastomas, small-cell lung carcinomas, and many sarcomas, while absent in most normal tissues. GD2 expression has been demonstrated in human melanoma and small cell lung cancer by thin layer chromatography and radiolabeled anti-GD2 antibody detection. It is hypothesized that one mode of action of MORAb-028 is complement-dependent cytotoxicity. Complement-dependent cytotoxicity is a mechanism for killing tumor cells in which an antibody bound to the target cell surface fixes complement, which results in assembly of the complement membrane attack complex that punches holes in the target cell membrane resulting in subsequent cell lysis. IgMs strongly bind to C1Q and robustly activate complement-dependent cytotoxicity. MORAb-028 is being developed as a potential therapy for GD2-positive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Measurable metastatic melanoma that has failed standard therapy
* Males and females greater than or equal to 18 years of age
* Life expectancy of greater than or equal to 3 months

Exclusion Criteria:

* Significant cardiovascular impairment
* Clinically significant illness, medical condition, surgical history, or laboratory abnormality that could affect the safety of the subject or negatively impact the study results
* Chemotherapy, radiotherapy, or immunotherapy within 3 weeks prior to administration to MORAb-028

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety of single dose radio labeled MORAb-028 in subjects with metastatic melanoma | Daily for 7 days followed by weekly for 2 weeks, then biweekly for 4 weeks

SECONDARY OUTCOMES:
Radiologic distribution of a single i.v. infusion of MORAb-028 | Daily for 1 week post study drug administration
Pharmacokinetic parameters of labeled and unlabeled MORAb-028 | Daily for 7 days followed by weekly for 2 weeks, then biweekly for 4 weeks
The incidence of human antihuman antibody formation | Week 2 and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Christina Coughlin, MD, PhD, Study Director — Morphotek; Jorge Carrasquillo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States